CLINICAL TRIAL: NCT03620032
Title: Phase 2 Randomized Study of RT and Reirradiation at Relapse vs Multiple Elective RT Courses With Same Concomitant CT for Newly Diagnosed
Brief Title: Study of Re-irradiation at Relapse Versus RT and Multiple Elective rt Courses
Acronym: DIPG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: University of Roma La Sapienza (Other); Johannes Gutenberg University Mainz (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-002185-23
Record Dates: First submitted 2018-05-14; First posted 2018-08-08 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Diffuse Intrinsic Pontine Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — nimotuzumab; Vinorelbine; Drug Therapy; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective, non-blinded, randomised two cohorts study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (Other): Nimotuzumab 150 mg /mq/d as iv weekly and Vinorelbine 20 mg/mq/d weekly, in week 1-12 (Induction phase).If not progression Nimotuzumab 150 mg/m2 as iv and Vinorelbine 25 mg/m²/d as iv until progression or maximum at week 108; in case of non-progressive disease re-irradiation 1 for a total of 19.8 Gy from week 26 to week 28; in case of non-progressive disease: re-irradiation 2 for a total of 19.8 Gy from week 46 to week 48. Irradiation will be scheduled to begin in the 3rd week after starting the nimotuzumab and vinorelbine treatment. For the first course, a total dose of 36 Gy will be delivered, in 1.8 Gy daily fractions 5 days a week.
  Interventions: Drug: Nimotuzumab; Drug: Vinorelbine; Other: Radiotherapy
- Experimental treatment (Experimental): Nimotuzumab 150 mg /mq/d as iv weekly and Vinorelbine 20 mg/mq/d weekly, in week 1-12 (Induction phase).If not progression Nimotuzumab 150 mg/m2 as iv and Vinorelbine 25 mg/m²/d as iv until progression or maximum at week 108; in case of non-progressive disease re-irradiation 1 for a total of 19.8 Gy from week 26 to week 28; in case of non-progressive disease: re-irradiation 2 for a total of 19.8 Gy from week 46 to week 48. Irradiation will be scheduled to begin in the 3rd week after starting the nimotuzumab and vinorelbine treatment. For the first course, a total dose of 36 Gy will be delivered, in 1.8 Gy daily fractions 5 days a week.
  Interventions: Drug: Nimotuzumab; Drug: Vinorelbine; Other: Radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — humanized therapeutic monoclonal antibody against epidermal growth factor receptor (EGFR)
  Other Names: humanized therapeutic monoclonal antibody
Drug: Vinorelbine — Chemotherapy
  Other Names: Chemotherapy
Other: Radiotherapy — RADIOTHERAPY SCHEDULE IS DESCRIBED FOR BOTH GROUPS IN THE PERAGRAPH TITLET ARMS

SUMMARY:
Prospective, non-blinded, randomised two cohorts study on the efficacy of two different radiotherapy schedule for DIPG by using the same concomitant and post-radiotherapy systemic treatment.

DETAILED DESCRIPTION:
1. st cohort: Standard Arm with Radiotherapy, Nimotuzumab and vinorelbine Nimotuzumab 150 mg /m2/d as iv short-term infusion for 30 min weekly in week 1-12 and Vinorelbine 20 mg/m2/d weekly in week 1-12 as iv short-term infusion for 30 min (Induction phase).1st re-evaluation week 13 (day 85-91). In case of non-progressive disease: Nimotuzumab 150 mg/m2/d iv short-term infusion for 30 min and Vinorelbine 25 mg/m2/d as iv short-term infusion for 30 min every two weeks in week 14, 16, 18, 20, 22, 24 (Consolidation phase I) 2nd re-evaluation week 25, thereafter in case of non-progressive disease.Nimotuzumab 150 mg/m2/d iv short-term infusion for 30 min and Vinorelbine 25 mg/m2/d as iv short-term infusion for 30 min every two weeks , with re-evaluation at week 37 and any 12 weeks until progression or maximum at week 108. Irradiation will be scheduled to begin in the 3rd week after starting the nimotuzumab and vinorelbine treatment. A total dose of 54 Gy will be delivered, in 1.8 Gy daily fractions 5 days a week, with a 6 MV linear accelerator. To plan radiotherapy, CT images will be acquired with a 2 mm slice thickness, with patients positioned ready for treatment, their heads immobilized with a custom-made thermoplastic mask. Each patient's CT images will be co-registered with T2-weighted, gadolinium enhanced T1-weighted, and fluid-attenuated inversion recovery MRI sequences to identify the gross target volume (GTV) precisely. A three-dimensional conformal radiotherapy technique with 5 or 6 coplanar or non-coplanar beams or an intensity modulated radiotherapy technique will be adopted.

   Re-irradiation at progression.In case of local progressive disease, after obtaining a new consent from parents/patient if the case, a full course of re-irradiation will be proposed with 19.8 Gy, fractionated over 11 days.
2. -cohort: Experimental arm with Nimotuzumab + Vinorelbine and refracted radiotherapy doses. Nimotuzumab 150 mg/m2/d as iv short-term infusion for 30 min weekly in week 1-12 and Vinorelbine weekly 20 mg/m2/d in week 1-12 as iv short-term infusion for 30 min (Induction phase, as for standard arm); 1st re-evaluation week 13. In case of non-progressive disease, any other week, Nimotuzumab 150 mg/m2 as iv short-term infusion for 30 min and Vinorelbine 25 mg/m2/d as iv short-term infusion for 30 min until progression or maximum at week 108;2nd re-evaluation week 25, thereafter in case of non-progressive disease re-irradiation one for a total of 19.8 Gy in 11 fractions at 1.8 Gy/day from week 26 to week 28 together with vinorelbine/nimotuzumab continuation any other week;3rd re-evaluation week 37, thereafter in case of non-progressive disease vinorelbine/nimotuzumab continuation any other week;4th re-evaluation week 45, thereafter in case of non-progressive disease: re-irradiation two for a total of 19.8 Gy in 11 fractions at 1.8 Gy/day from week 46 to week 48 together with vinorelbine/nimotuzumab continuation any other week;Further re-evaluation will be done at week 61 and thereafter any 12 weeks as for standard arm continuing vinorelbine and nimotuzumab until progression or maximum at week 108 .Patients will continue with re-irradiation courses also in case of progressive disease, and will continue to be evaluated for OS.Irradiation will be scheduled to begin in the 3rd week after starting the nimotuzumab and vinorelbine treatment. For the first course, a total dose of 36 Gy will be delivered, in 1.8 Gy daily fractions 5 days a week, with a 6 MV linear accelerator. To plan radiotherapy, CT images will be acquired with a 2 mm slice thickness, with patients positioned ready for treatment, their heads immobilized with a custom-made thermoplastic mask. Each patient's CT images will be co-registered with T2-weighted, gadolinium enhanced T1-weighted, and fluid-attenuated inversion recovery MRI sequences to identify the gross target volume (GTV) precisely. A three-dimensional conformal radiotherapy technique with 5 or 6 coplanar or non-coplanar beams or an intensity modulated radiotherapy technique will be adopted.The second course will be planned after second evaluation. It will be scheduled from week 26 to week 28 and planning will follow same guidelines as first course. The course of re-irradiation will be proposed with 19.8 Gy, fractionated over 11 days.

The third and last course will be planned after forth evaluation. It will be scheduled from week 46 to week 48 and planning will follow same guidelines as first and second course (radiation and first re-irradiation). The course of re-irradiation will be proposed with 19.8 Gy, fractionated over 11 days.

Re-irradiation at progression. n case of local progressive disease after the whole three radiotherapy courses, after obtaining a new consent form parents/patient if the case, a course of re-irradiation will be proposed with 9 Gy total dose, fractionated over 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 2 to 21 years old will be eligible
* No previous treatment consented apart from steroids
* Strict eligibility criteria will radiologically-verified DIPG (an intrinsic, pontine-based infiltrative lesion hypointense on T1- and hyperintense on T2-weighted sequences, involving at least 2/3 of the pons)
* symptoms lasting less than 6 months, life expectancy ≥4 weeks; Karnowski/Lansky performance status ≥ 40 %
* no organ dysfunction; no pregnancy or breast-feeding
* Patients undergo baseline cranial MRI with gadolinium, to be repeated if treatment begins more than 2 weeks; spinal MRI due to the occurrence of metastatic cases at diagnosis will also be mandatory
* Written and signed informed consent from parents or legal guardians will be obtained before starting the treatment.

Exclusion Criteria:

* Patients below 2 years or over 21
* Pre-treatment with radio or chemotherapy
* Neurofibromatosis 1
* Non-typical imaging
* Symptoms duration over 6 months, Lansky/Karnowski scores below 40%
* Metastatic disease as shown by MRI
* Organ dysfunction, pregnancy or breast-feeding
* Absence of parents, patient or tutor consent

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2024-11-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 years
  Primary aim of this study will be to compare the best response up to 36 weeks (CR+PR) between conventional and experimental irradiation. Such an end point was chosen since tumor reduction has been demonstrated to be correlated with better PFS and OS. The response will be evaluated according to radiological and clinical criteria. Radiological criteria will be RECIST ones.

SECONDARY OUTCOMES:
disease stabilization rate | 3 years
  the disease stabilization rates (considering only the number of patients with stable disease) will be calculated in the two treatment arms, together with the corresponding binomial 95% confidence intervals.
PFS | 3 years
  Progression-free survival (PFS) will be measured from the date of randomisation to the date of event, defined as progression or death due to any cause. Patients with no event as the time of the analysis will be censored at their last adequate tumour assessment. PFS will be estimated in the two treatment arms by the Kaplan-Meier method.
OS | 3 years
  Overall survival (OS) will be measured from the date of randomisation to the date of death due to any cause and will be censored at the date of last follow-up for patients alive at their last follow-up. OS will be estimated in the two treatment arms by the Kaplan-Meier method.
radiotherapy toxicity (adverse events) | 3 years
  The toxicity will be measured through the control of adverse events. The evaluation of adverse events will be done through the CTCAE 4.03 table.
PedsQL (Paediatric Quality of Life Questionnaire) | 3 years
  quality of life evaluation;
EORTC QLQ-C30 (Quality of Life Questionnaire) | 3 years
  quality of life evaluation
Brain module (BN20) | 3 years
  quality of life evaluation
SDQ (Strength and Difficulties Questionnaire) | 3 years
  quality of life evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Maura Massimino, MD, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bode U, Buchen S, Warmuth-Metz M, Pietsch T, Bach F, Fleischhack G. Final report of a phase II trial of nimotuzumab in the treatment of refractory and relapsed high-grade gliomas in children and adolescents [abstract]. J Clin Oncol (2007); 25(Suppl. 2006)
- [Result] Bartels U, Wolff J, Gore L, Dunkel I, Gilheeney S, Allen J, Goldman S, Yalon M, Packer RJ, Korones DN, Smith A, Cohen K, Kuttesch J, Strother D, Baruchel S, Gammon J, Kowalski M, Bouffet E. Phase 2 study of safety and efficacy of nimotuzumab in pediatric patients with progressive diffuse intrinsic pontine glioma. Neuro Oncol. 2014 Nov;16(11):1554-9. doi: 10.1093/neuonc/nou091. Epub 2014 May 20. PMID 24847085
- [Result] Bernier-Chastagner V, Grill J, Doz F, Bracard S, Gentet JC, Marie-Cardine A, Luporsi E, Margueritte G, Lejars O, Laithier V, Mechinaud F, Millot F, Kalifa C, Chastagner P. Topotecan as a radiosensitizer in the treatment of children with malignant diffuse brainstem gliomas: results of a French Society of Paediatric Oncology Phase II Study. Cancer. 2005 Dec 15;104(12):2792-7. doi: 10.1002/cncr.21534. PMID 16265674
- [Result] Bode U, Massimino M, Bach F, Zimmermann M, Khuhlaeva E, Westphal M, Fleischhack G. Nimotuzumab treatment of malignant gliomas. Expert Opin Biol Ther. 2012 Dec;12(12):1649-59. doi: 10.1517/14712598.2012.733367. Epub 2012 Oct 8. PMID 23043252
- [Result] Clerk-Lamalice O, Reddick WE, Li X, Li Y, Edwards A, Glass JO, Patay Z. MRI Evaluation of Non-Necrotic T2-Hyperintense Foci in Pediatric Diffuse Intrinsic Pontine Glioma. AJNR Am J Neuroradiol. 2016 Oct;37(10):1930-1937. doi: 10.3174/ajnr.A4814. Epub 2016 May 19. PMID 27197987
- [Result] Conway AE, Reddick WE, Li Y, Yuan Y, Glass JO, Baker JN, Kun LE, Broniscer A, Patay Z. "Occult" post-contrast signal enhancement in pediatric diffuse intrinsic pontine glioma is the MRI marker of angiogenesis? Neuroradiology. 2014 May;56(5):405-12. doi: 10.1007/s00234-014-1348-9. Epub 2014 Mar 14. PMID 24626721
- [Result] Lobel U, Sedlacik J, Reddick WE, Kocak M, Ji Q, Broniscer A, Hillenbrand CM, Patay Z. Quantitative diffusion-weighted and dynamic susceptibility-weighted contrast-enhanced perfusion MR imaging analysis of T2 hypointense lesion components in pediatric diffuse intrinsic pontine glioma. AJNR Am J Neuroradiol. 2011 Feb;32(2):315-22. doi: 10.3174/ajnr.A2277. Epub 2010 Nov 18. PMID 21087935
- [Result] Hargrave D, Chuang N, Bouffet E. Conventional MRI cannot predict survival in childhood diffuse intrinsic pontine glioma. J Neurooncol. 2008 Feb;86(3):313-9. doi: 10.1007/s11060-007-9473-5. Epub 2007 Oct 2. PMID 17909941
- [Result] Jansen MH, Veldhuijzen van Zanten SE, Sanchez Aliaga E, Heymans MW, Warmuth-Metz M, Hargrave D, van der Hoeven EJ, Gidding CE, de Bont ES, Eshghi OS, Reddingius R, Peeters CM, Schouten-van Meeteren AY, Gooskens RH, Granzen B, Paardekooper GM, Janssens GO, Noske DP, Barkhof F, Kramm CM, Vandertop WP, Kaspers GJ, van Vuurden DG. Survival prediction model of children with diffuse intrinsic pontine glioma based on clinical and radiological criteria. Neuro Oncol. 2015 Jan;17(1):160-6. doi: 10.1093/neuonc/nou104. Epub 2014 Jun 5. PMID 24903904
- [Result] Poussaint TY, Kocak M, Vajapeyam S, Packer RI, Robertson RL, Geyer R, Haas-Kogan D, Pollack IF, Vezina G, Zimmerman R, Cha S, Patay Z, Boyett JM, Kun LE. MRI as a central component of clinical trials analysis in brainstem glioma: a report from the Pediatric Brain Tumor Consortium (PBTC). Neuro Oncol. 2011 Apr;13(4):417-27. doi: 10.1093/neuonc/noq200. Epub 2011 Feb 4. PMID 21297126
- [Result] Zaghloul MS, Eldebawy E, Ahmed S, Mousa AG, Amin A, Refaat A, Zaky I, Elkhateeb N, Sabry M. Hypofractionated conformal radiotherapy for pediatric diffuse intrinsic pontine glioma (DIPG): a randomized controlled trial. Radiother Oncol. 2014 Apr;111(1):35-40. doi: 10.1016/j.radonc.2014.01.013. Epub 2014 Feb 20. PMID 24560760
- [Result] Wolff JE, Westphal S, Molenkamp G, Gnekow A, Warmuth-Metz M, Rating D, Kuehl J. Treatment of paediatric pontine glioma with oral trophosphamide and etoposide. Br J Cancer. 2002 Oct 21;87(9):945-9. doi: 10.1038/sj.bjc.6600552. PMID 12434281
- [Result] Wolff JE, Wagner S, Reinert C, Gnekow A, Kortmann RD, Kuhl J, Van Gool SW. Maintenance treatment with interferon-gamma and low-dose cyclophosphamide for pediatric high-grade glioma. J Neurooncol. 2006 Sep;79(3):315-21. doi: 10.1007/s11060-006-9147-8. Epub 2006 Apr 28. PMID 16645718
- [Result] Wolff JE, Kortmann RD, Wolff B, Pietsch T, Peters O, Schmid HJ, Rutkowski S, Warmuth-Metz M, Kramm C. High dose methotrexate for pediatric high grade glioma: results of the HIT-GBM-D pilot study. J Neurooncol. 2011 May;102(3):433-42. doi: 10.1007/s11060-010-0334-2. Epub 2010 Aug 8. PMID 20694800
- [Result] Wolff JE, Driever PH, Erdlenbruch B, Kortmann RD, Rutkowski S, Pietsch T, Parker C, Metz MW, Gnekow A, Kramm CM. Intensive chemotherapy improves survival in pediatric high-grade glioma after gross total resection: results of the HIT-GBM-C protocol. Cancer. 2010 Feb 1;116(3):705-12. doi: 10.1002/cncr.24730. PMID 19957326
- [Result] Wagner S, Warmuth-Metz M, Emser A, Gnekow AK, Strater R, Rutkowski S, Jorch N, Schmid HJ, Berthold F, Graf N, Kortmann RD, Pietsch T, Sorensen N, Peters O, Wolff JE. Treatment options in childhood pontine gliomas. J Neurooncol. 2006 Sep;79(3):281-7. doi: 10.1007/s11060-006-9133-1. Epub 2006 Apr 6. PMID 16598416
- [Result] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Result] Sufit A, Donson AM, Birks DK, Knipstein JA, Fenton LZ, Jedlicka P, Hankinson TC, Handler MH, Foreman NK. Diffuse intrinsic pontine tumors: a study of primitive neuroectodermal tumors versus the more common diffuse intrinsic pontine gliomas. J Neurosurg Pediatr. 2012 Aug;10(2):81-8. doi: 10.3171/2012.3.PEDS11316. Epub 2012 Jun 29. PMID 22747092
- [Result] Bogaerts J, Sydes MR, Keat N, McConnell A, Benson A, Ho A, Roth A, Fortpied C, Eng C, Peckitt C, Coens C, Pettaway C, Arnold D, Hall E, Marshall E, Sclafani F, Hatcher H, Earl H, Ray-Coquard I, Paul J, Blay JY, Whelan J, Panageas K, Wheatley K, Harrington K, Licitra L, Billingham L, Hensley M, McCabe M, Patel PM, Carvajal R, Wilson R, Glynne-Jones R, McWilliams R, Leyvraz S, Rao S, Nicholson S, Filiaci V, Negrouk A, Lacombe D, Dupont E, Pauporte I, Welch JJ, Law K, Trimble T, Seymour M. Clinical trial designs for rare diseases: studies developed and discussed by the International Rare Cancers Initiative. Eur J Cancer. 2015 Feb;51(3):271-81. doi: 10.1016/j.ejca.2014.10.027. Epub 2014 Dec 24. PMID 25542058
- [Result] Chen K, Shan M. Optimal and minimax three-stage designs for phase II oncology clinical trials. Contemp Clin Trials. 2008 Jan;29(1):32-41. doi: 10.1016/j.cct.2007.04.008. Epub 2007 May 6. PMID 17544337
- [Result] Rutka JT. Biopsy of diffuse intrinsic pontine gliomas? J Neurosurg Pediatr. 2012 Aug;10(2):79-80. doi: 10.3171/2012.2.PEDS1237. Epub 2012 Jun 29. No abstract available. PMID 22747087
- [Result] Roujeau T, Machado G, Garnett MR, Miquel C, Puget S, Geoerger B, Grill J, Boddaert N, Di Rocco F, Zerah M, Sainte-Rose C. Stereotactic biopsy of diffuse pontine lesions in children. J Neurosurg. 2007 Jul;107(1 Suppl):1-4. doi: 10.3171/PED-07/07/001. PMID 17647306
- [Result] Pollack IF, Stewart CF, Kocak M, Poussaint TY, Broniscer A, Banerjee A, Douglas JG, Kun LE, Boyett JM, Geyer JR. A phase II study of gefitinib and irradiation in children with newly diagnosed brainstem gliomas: a report from the Pediatric Brain Tumor Consortium. Neuro Oncol. 2011 Mar;13(3):290-7. doi: 10.1093/neuonc/noq199. Epub 2011 Feb 3. PMID 21292687
- [Result] Packer RJ, Krailo M, Mehta M, Warren K, Allen J, Jakacki R, Villablanca JG, Chiba A, Reaman G. Phase 1 study of concurrent RMP-7 and carboplatin with radiotherapy for children with newly diagnosed brainstem gliomas. Cancer. 2005 Sep 15;104(6):1281-7. doi: 10.1002/cncr.21301. PMID 16078267
- [Result] Negretti L, Bouchireb K, Levy-Piedbois C, Habrand JL, Dhermain F, Kalifa C, Grill J, Dufour C. Hypofractionated radiotherapy in the treatment of diffuse intrinsic pontine glioma in children: a single institution's experience. J Neurooncol. 2011 Sep;104(3):773-7. doi: 10.1007/s11060-011-0542-4. Epub 2011 Feb 17. PMID 21327862
- [Result] Massimino M, Spreafico F, Biassoni V, Simonetti F, Riva D, Trecate G, Giombini S, Poggi G, Pecori E, Pignoli E, Casanova M, Ferrari A, Meazza C, Luksch R, Terenziani M, Cefalo G, Podda M, Polastri D, Clerici CA, Fossati-Bellani F, Gandola L. Diffuse pontine gliomas in children: changing strategies, changing results? A mono-institutional 20-year experience. J Neurooncol. 2008 May;87(3):355-61. doi: 10.1007/s11060-008-9525-5. Epub 2008 Jan 24. PMID 18217208
- [Result] Massimino M, Bode U, Biassoni V, Fleischhack G. Nimotuzumab for pediatric diffuse intrinsic pontine gliomas. Expert Opin Biol Ther. 2011 Feb;11(2):247-56. doi: 10.1517/14712598.2011.546341. Epub 2010 Dec 21. PMID 21171927
- [Result] Massimino M, Biassoni V, Miceli R, Schiavello E, Warmuth-Metz M, Modena P, Casanova M, Pecori E, Giangaspero F, Antonelli M, Buttarelli FR, Potepan P, Pollo B, Nunziata R, Spreafico F, Podda M, Anichini A, Clerici CA, Sardi I, De Cecco L, Bode U, Bach F, Gandola L. Results of nimotuzumab and vinorelbine, radiation and re-irradiation for diffuse pontine glioma in childhood. J Neurooncol. 2014 Jun;118(2):305-312. doi: 10.1007/s11060-014-1428-z. Epub 2014 Apr 3. PMID 24696052
- [Result] MacDonald TJ. Diffuse intrinsic pontine glioma (DIPG): time to biopsy again? Pediatr Blood Cancer. 2012 Apr;58(4):487-8. doi: 10.1002/pbc.24090. No abstract available. PMID 22331797
- [Result] Lassman LP, Arjona VE. Pontine gliomas of childhood. Lancet. 1967 Apr 29;1(7496):913-5. doi: 10.1016/s0140-6736(67)91485-7. No abstract available. PMID 4164397
- [Result] Kretschmar CS, Tarbell NJ, Barnes PD, Krischer JP, Burger PC, Kun L. Pre-irradiation chemotherapy and hyperfractionated radiation therapy 66 Gy for children with brain stem tumors. A phase II study of the Pediatric Oncology Group, Protocol 8833. Cancer. 1993 Aug 15;72(4):1404-13. doi: 10.1002/1097-0142(19930815)72:43.0.co;2-g. PMID 8339231
- [Result] Jennings MT, Sposto R, Boyett JM, Vezina LG, Holmes E, Berger MS, Bruggers CS, Bruner JM, Chan KW, Dusenbery KE, Ettinger LJ, Fitz CR, Lafond D, Mandelbaum DE, Massey V, McGuire W, McNeely L, Moulton T, Pollack IF, Shen V. Preradiation chemotherapy in primary high-risk brainstem tumors: phase II study CCG-9941 of the Children's Cancer Group. J Clin Oncol. 2002 Aug 15;20(16):3431-7. doi: 10.1200/JCO.2002.04.109. PMID 12177103
- [Result] Jennings MT, Freeman ML, Murray MJ. Strategies in the treatment of diffuse pontine gliomas: the therapeutic role of hyperfractionated radiotherapy and chemotherapy. J Neurooncol. 1996 May-Jun;28(2-3):207-22. doi: 10.1007/BF00250200. PMID 8832463
- [Result] Janssens GO, Gidding CE, Van Lindert EJ, Oldenburger FR, Erasmus CE, Schouten-Meeteren AY, Kaanders JH. The role of hypofractionation radiotherapy for diffuse intrinsic brainstem glioma in children: a pilot study. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):722-6. doi: 10.1016/j.ijrobp.2008.05.030. Epub 2008 Nov 5. PMID 18990510
- [Result] Jackson S, Patay Z, Howarth R, Pai Panandiker AS, Onar-Thomas A, Gajjar A, Broniscer A. Clinico-radiologic characteristics of long-term survivors of diffuse intrinsic pontine glioma. J Neurooncol. 2013 Sep;114(3):339-44. doi: 10.1007/s11060-013-1189-0. Epub 2013 Jun 29. PMID 23813229
- [Result] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Result] Harris W. A Case of Pontine Glioma, with Special Reference to the Paths of Gustatory Sensation. Proc R Soc Med. 1926;19(Neurol Sect):1-5. doi: 10.1177/003591572601900901. No abstract available. PMID 19985059
- [Result] Hargrave D, Bartels U, Bouffet E. Diffuse brainstem glioma in children: critical review of clinical trials. Lancet Oncol. 2006 Mar;7(3):241-8. doi: 10.1016/S1470-2045(06)70615-5. PMID 16510333
- [Result] Gilbertson RJ, Hill DA, Hernan R, Kocak M, Geyer R, Olson J, Gajjar A, Rush L, Hamilton RL, Finkelstein SD, Pollack IF. ERBB1 is amplified and overexpressed in high-grade diffusely infiltrative pediatric brain stem glioma. Clin Cancer Res. 2003 Sep 1;9(10 Pt 1):3620-4. PMID 14506149
- [Result] Geyer JR, Stewart CF, Kocak M, Broniscer A, Phillips P, Douglas JG, Blaney SM, Packer RJ, Gururangan S, Banerjee A, Kieran MW, Kun LE, Gilbertson RJ, Boyett JM. A phase I and biology study of gefitinib and radiation in children with newly diagnosed brain stem gliomas or supratentorial malignant gliomas. Eur J Cancer. 2010 Dec;46(18):3287-93. doi: 10.1016/j.ejca.2010.07.005. Epub 2010 Aug 12. PMID 20708924
- [Result] Geoerger B, Hargrave D, Thomas F, Ndiaye A, Frappaz D, Andreiuolo F, Varlet P, Aerts I, Riccardi R, Jaspan T, Chatelut E, Le Deley MC, Paoletti X, Saint-Rose C, Leblond P, Morland B, Gentet JC, Meresse V, Vassal G; ITCC (Innovative Therapies for Children with Cancer) European Consortium. Innovative Therapies for Children with Cancer pediatric phase I study of erlotinib in brainstem glioma and relapsing/refractory brain tumors. Neuro Oncol. 2011 Jan;13(1):109-18. doi: 10.1093/neuonc/noq141. Epub 2010 Oct 25. PMID 20974795
- [Result] Freeman CR, Farmer JP. Pediatric brain stem gliomas: a review. Int J Radiat Oncol Biol Phys. 1998 Jan 15;40(2):265-71. doi: 10.1016/s0360-3016(97)00572-5. PMID 9457808
- [Result] Frappaz D, Schell M, Thiesse P, Marec-Berard P, Mottolese C, Perol D, Bergeron C, Philip T, Ricci AC, Galand-Desme S, Szathmari A, Carrie C. Preradiation chemotherapy may improve survival in pediatric diffuse intrinsic brainstem gliomas: final results of BSG 98 prospective trial. Neuro Oncol. 2008 Aug;10(4):599-607. doi: 10.1215/15228517-2008-029. Epub 2008 Jun 24. PMID 18577561
- [Result] Fontanilla HP, Pinnix CC, Ketonen LM, Woo SY, Vats TS, Rytting ME, Wolff JE, Mahajan A. Palliative reirradiation for progressive diffuse intrinsic pontine glioma. Am J Clin Oncol. 2012 Feb;35(1):51-7. doi: 10.1097/COC.0b013e318201a2b7. PMID 21297433
- [Result] Feshchenko EA, Langdon WY, Tsygankov AY. Fyn, Yes, and Syk phosphorylation sites in c-Cbl map to the same tyrosine residues that become phosphorylated in activated T cells. J Biol Chem. 1998 Apr 3;273(14):8323-31. doi: 10.1074/jbc.273.14.8323. PMID 9525940
- [Result] Doz F, Neuenschwander S, Bouffet E, Gentet JC, Schneider P, Kalifa C, Mechinaud F, Chastagner P, De Lumley L, Sariban E, Plantaz D, Mosseri V, Bours D, Alapetite C, Zucker JM. Carboplatin before and during radiation therapy for the treatment of malignant brain stem tumours: a study by the Societe Francaise d'Oncologie Pediatrique. Eur J Cancer. 2002 Apr;38(6):815-9. doi: 10.1016/s0959-8049(02)00029-1. PMID 11937316
- [Result] Bradley KA, Zhou T, McNall-Knapp RY, Jakacki RI, Levy AS, Vezina G, Pollack IF. Motexafin-gadolinium and involved field radiation therapy for intrinsic pontine glioma of childhood: a children's oncology group phase 2 study. Int J Radiat Oncol Biol Phys. 2013 Jan 1;85(1):e55-60. doi: 10.1016/j.ijrobp.2012.09.004. Epub 2012 Oct 22. PMID 23092726
- [Result] Broniscer A, Baker JN, Tagen M, Onar-Thomas A, Gilbertson RJ, Davidoff AM, Pai Panandiker AS, Leung W, Chin TK, Stewart CF, Kocak M, Rowland C, Merchant TE, Kaste SC, Gajjar A. Phase I study of vandetanib during and after radiotherapy in children with diffuse intrinsic pontine glioma. J Clin Oncol. 2010 Nov 1;28(31):4762-8. doi: 10.1200/JCO.2010.30.3545. Epub 2010 Oct 4. PMID 20921456
- [Result] Broniscer A, Baker SJ, Stewart CF, Merchant TE, Laningham FH, Schaiquevich P, Kocak M, Morris EB, Endersby R, Ellison DW, Gajjar A. Phase I and pharmacokinetic studies of erlotinib administered concurrently with radiotherapy for children, adolescents, and young adults with high-grade glioma. Clin Cancer Res. 2009 Jan 15;15(2):701-7. doi: 10.1158/1078-0432.CCR-08-1923. PMID 19147777
- [Result] Boop FA. Brainstem gliomas. J Neurosurg Pediatr. 2011 Dec;8(6):537-8; discussion 538. doi: 10.3171/2011.8.PEDS11310. No abstract available. PMID 22132908
- [Result] Memorial Sloan-Kettering Cancer Center. External beam radiation therapy and cetuximab followed by irinotecan and cetuximab for children and young adults with newly diagnosed diffuse pontine tumors and high-grade astrocytomas (POE08-01). ClinicalTrials. gov identifier NCT01012609
- [Result] Fleischhack G, Siegler N, Zimmermann M, et al. Concomitant therapy of nimotuzumab and standard radiotherapy for the treatment of newly diagnosed diffuse intrinsic pontine gliomas in children and adolescents. 14th international symposium of pediatric neuro-oncology, Vienna, Austria 20-23 June 2010
- [Result] Broniscer A, Baker SD, Wetmore C, Pai Panandiker AS, Huang J, Davidoff AM, Onar-Thomas A, Panetta JC, Chin TK, Merchant TE, Baker JN, Kaste SC, Gajjar A, Stewart CF. Phase I trial, pharmacokinetics, and pharmacodynamics of vandetanib and dasatinib in children with newly diagnosed diffuse intrinsic pontine glioma. Clin Cancer Res. 2013 Jun 1;19(11):3050-8. doi: 10.1158/1078-0432.CCR-13-0306. Epub 2013 Mar 27. PMID 23536435